CLINICAL TRIAL: NCT04578873
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled, Ascending Single- and Multiple-Dose Study of the Safety, Tolerability, and Pharmacokinetics of Oral QPX7831 in Healthy Adult Subjects
Brief Title: Phase 1 Oral QPX7831 SAD and MAD in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Qpex Biopharma, Inc. (Industry)
Collaborators: Biomedical Advanced Research and Development Authority (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Qpex-101
Record Dates: First submitted 2020-09-29; First posted 2020-10-08 (Actual); Last update posted 2022-10-10 (Actual); Status verified 2022-09

CONDITIONS: Bacterial Infections
Keywords: beta-lactamase inhibitor
MeSH Terms: conditions — Bacterial Infections

STUDY DESIGN:
Intervention Model Description: Double-blind, placebo-controlled, sequential, ascending single-and multiple-dose design
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: matched oral placebo capsule
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- QPX7831 SAD Cohorts (Experimental): oral, single ascending dose (or placebo)
  Interventions: Drug: QPX7831; Drug: placebo comparator
- QPX7831 MAD Cohorts (Experimental): oral, multiple ascending dose (or placebo)
  Interventions: Drug: QPX7831; Drug: placebo comparator

INTERVENTIONS:
Drug: QPX7831 — capsule
Drug: placebo comparator — oral matched placebo capsule

SUMMARY:
This Phase 1 study will assess the safety, tolerability, and pharmacokinetics (PK) of QPX7831, a beta-lactamase inhibitor, when administered orally in single ascending doses and in multiple ascending doses to heathy adult subjects.

DETAILED DESCRIPTION:
Qpex Biopharma, Inc. is developing an oral dosage form that delivers QPX7728, a new boron-based beta-lactamase inhibitor with activity against both serine and metallo-beta-lactamases, for oral treatment in combination with a beta-lactam antibiotic.

The objectives are:

1. To assess the safety and tolerability of QPX7831 when administered orally in single ascending doses (SAD) and in multiple ascending doses (MAD) to healthy adult subjects.
2. To assess the PK of single and multiple doses of oral QPX7831 when administered to healthy adult subjects to determine if the target exposures identified in preclinical studies can be attained in healthy adult subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult males and/or females of non-childbearing potential, 18 to 55 years of age (inclusive) at the time of screening.
2. Body mass index (BMI) ≥ 18.5 and ≤ 29.9 (kg/m2) and weight between 55.0 and 100.0 kg (inclusive).
3. Medically healthy with clinically insignificant screening results (e.g., laboratory profiles, medical histories, electrocardiograms [ECGs], physical examination) as assessed by the PI.
4. Voluntarily consent to participate in the study.
5. Male volunteers must agree to use a condom when engaging in any sexual activity from study check-in through 30 days following the last administration of the study drug, and to not donate sperm during this same period of time. If engaging in sexual activity with a female partner of childbearing potential, an additional method of birth control must be used. Approved additional methods of birth control include:

   1. Intra-uterine device (IUD) in place for at least 3 months prior to Day 1 through 30 days following the final dosing of the study drug.
   2. Barrier method (diaphragm) for at least 14 days prior to Day 1 through 30 days following dosing of the study drug.
   3. Stable hormonal contraceptive for at least 3 months prior to Day 1 through 30 days following dosing of the study drug.
   4. Surgical sterilization (vasectomy) at least 6 months prior to Day 1.
6. Females of non-childbearing potential with serum FSH levels ≥ 40 mIU/mL are either postmenopausal (defined as 12 months spontaneous amenorrhea) or have undergone one of the following sterilization procedures at least 6 months prior to Day 1 (and is documented):

   1. Bilateral tubal ligation;
   2. Hysterectomy;
   3. Hysterectomy with unilateral or bilateral oophorectomy;
   4. Bilateral oophorectomy.

Exclusion Criteria:

1. History or presence of significant cardiovascular, pulmonary, hepatic, renal, hematological, gastrointestinal, endocrine, immunologic, dermatologic, neurological, or psychiatric disease.
2. Positive urine drug/alcohol testing at screening or check-in (Day -1).
3. Positive testing for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), or hepatitis C antibodies (HCV).
4. History or presence of alcoholism or drug abuse within the 2 years prior to Day 1.
5. Use of more than 5 packs/week of cigarettes (or equivalent amount of nicotine-containing product) within 6 months prior to Day 1. Subjects must agree to refrain from smoking for the duration of the study.
6. Excessive intake of alcohol, defined as an average daily intake of greater than 2 standard drinks for women and 4 standard drinks for men; 1 bottle of beer (375mL) is equivalent to approximately 1.4 standard drinks, 1 glass of spirits (30mL) is equivalent to approximately 1 standard drink and 1 glass (150mL) of wine is equivalent to approximately 1.5 standard drinks.
7. Use of any prescription medication (with the exception of hormone replacement therapy for females) within 14 days prior to Day 1.
8. Use of any over the counter (OTC) medication, including herbal products, probiotics and vitamins, within the 7 days prior to Day 1. Up to 2 grams per day of paracetamol is allowed for acute events at the discretion of the PI.
9. Use of antacids, H2 receptor blockers or proton pump inhibitors within 7 days prior to Day 1.
10. Documented hypersensitivity reaction or anaphylaxis to any medication
11. Blood donation or significant blood loss (i.e., > 500 mL) within 56 days prior to Day
12. Plasma donation within 7 days prior to Day 1.
13. Participation in another investigational clinical trial within 30 days prior to Day 1 or within 5 half-lives of the previous investigational drug, whichever is longer.
14. Females who are pregnant or lactating.
15. Surgery within the past three months prior to Day 1 determined by the PI to be clinically relevant.
16. Any acute illness within 30 days prior to Day 1.
17. QTcF interval >450 msec for males and >470 for females or history of prolonged QT syndrome at screening or check-in (Day -1).
18. Calculated creatinine clearance less than 80 mL/min (Cockcroft-Gault method) at screening or check-in (Day -1).
19. Subjects who have any clinically significant abnormalities on laboratory values at screening or check-in (Day -1), in particular:

    1. White blood cell count < 3,000/mm3, hemoglobin < 11g/dL.
    2. Absolute neutrophil count < 1,200/mm3 or platelet count < 120,000/mm3.
    3. Liver function abnormalities at screening or check-in (Day -1) (defined by an elevation in bilirubin, AST or ALT 1.5 x ULN of the normal range for subjects based on age and sex).
20. Any other condition or prior therapy, which, in the opinion of the PI, would make the subject unsuitable for this study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2021-04-13 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2022-08-30 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment -Emergent Adverse events by subject and by cohort (single dose, multiple doses) | up to 17 days
  Number of patients with Treatment-Emergent AEs by subject, by cohort, severity and relationship to treatment
Number of patients with changes from baseline in safety parameters | up to 17 days
  Number of patients with changes in safety parameters before and after dosing by subject and cohort
Peak plasma Concentration measurements by subject and by cohort (Cmax) | up to 17 days
  Comparison will be performed between the cohorts for Cmax. Mean graphical presentation of the data will be reported. Statistical analysis of exposure parameters will be performed.
Time concentration data measurements by subject and by cohort (Tmax) | up to 17 days
  Comparison will be performed between the cohorts for Tmax.
Area under the plasma concentration versus time curve (AUC) between cohorts | up to 17 days
  Comparison will be performed between the cohorts for AUC. Mean graphical presentation of the data will be reported. Statistical analysis of exposure parameters will be performed.
Urine PK amount excreted by subject and by cohort | up to 17 days
  Urine PK parameters such as amount excreted will be calculated from urinary excretion data
Urine PK % dose excreted by subject and by cohort | up to 17 days
  Urine PK parameters such as amount of % dose excreted will be calculated from urinary excretion data

CONTACTS AND LOCATIONS:
Overall Officials: Jeffery Loutit, MBChB, Study Director — Qpex Biopharma, Inc.
Locations (2):
- Altasciences, Cypress, California, United States
- CMAX, Adelaide, South Australia, Australia

IPD SHARING:
Plan to Share IPD: No